CLINICAL TRIAL: NCT02153333
Title: Blinded Retrospective Laboratory Evaluations to Assess the Serologic Response to Porcine Circovirus Type 1 (PCV-1) in Infants Following the Administration of GlaxoSmithKline (GSK) Biologicals' Human Rotavirus Vaccine (444563)
Brief Title: Serologic Response to Porcine Circovirus Type 1 (PCV-1) in Infants Following Administration of Rotarix™
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114793; 444563/005 (Rota-005); 444563/023 (Rota-023); 444563/028 (Rota-028); 444563/029 (Rota-029); 102247 (Rota-036); 106481 (Rota-054)
Record Dates: First submitted 2014-05-15; First posted 2014-06-03 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Rotavirus
Keywords: Human rotavirus (HRV) vaccine; Serologic response; Porcine circovirus type 1 (PCV-1); Laboratory evaluations
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum samples

GROUPS / COHORTS (2):
- HRV Group: Subjects who had received 2 doses of HRV vaccine in previous studies.
  Interventions: Procedure: Serum sample
- Placebo Group: Subjects who had received 2 doses of placebo in previous studies.
  Interventions: Procedure: Serum sample

INTERVENTIONS:
Procedure: Serum sample — Serum samples collected at pre-vaccination and at 1-2 months post Dose 2 in the previously conducted clinical trials will be assessed for anti-PCV-1 antibodies in this study. Additionally, pre-vaccination sera samples from any infants testing positive for PCV-1 antibodies at the post-vaccination time point will also be evaluated.

SUMMARY:
This study aims to evaluate the serologic response to PCV-1 in the serum samples previously collected during initiation of vaccination series of Human Rotavirus (HRV) vaccine studies (1-2 months post Dose 2 of HRV vaccine or placebo). Additionally, pre-vaccination sera samples from any infants testing positive for PCV-1 antibodies at the post-vaccination time point will also be evaluated.

DETAILED DESCRIPTION:
Serum samples collected from 6 clinical trials previously conducted for HRV vaccine (Rotarix™) are used in this study.

ELIGIBILITY:
Inclusion Criteria:

Not applicable as no subjects will be actively enrolled in this study, only the sera samples of the subjects who were a part of previously conducted trials will be used for testing. However, the archived serum samples of only those subjects who satisfy the following criteria will be included in this study:

* Subjects who received two doses of HRV vaccine or Placebo and were included in the ATP cohort for immunogenicity in the primary studies listed.
* Subjects for whom their parents or Legally Acceptable Representatives (LARs) had agreed that their child or wards blood samples could be used for further research while giving consent for any of the primary studies listed.
* Subjects who have sufficient residual volume of serum samples at both pre- and post-vaccination time points.

Exclusion Criteria:

* Not Applicable

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged 6 to 12 weeks from 6 previously completed clinical trials, who received 2 doses of either Rotarix™ or Placebo.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Seropositivity rates for anti-PCV-1 antibodies. | At 1-2 months post dose 2 of HRV vaccine or placebo.
Seroconversion rates for anti-PCV-1 antibodies. | At 1-2 months post dose 2 of HRV vaccine or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Han HH, Karkada N, Jayadeva G, Dubin G. Serologic response to porcine circovirus type 1 (PCV1) in infants vaccinated with the human rotavirus vaccine, Rotarix: A retrospective laboratory analysis. Hum Vaccin Immunother. 2017 Jan 2;13(1):237-244. doi: 10.1080/21645515.2016.1231262. PMID 27657348